CLINICAL TRIAL: NCT01430728
Title: Cerebral Tissue Oxygen Saturation in Preterm Neonates Below 1500g Birth Weight During the First 72 Hours
Brief Title: Cerebral Tissue Oxygenation in Very Low Birthweight Infants in the First 3 Days of Life
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Manuel Schmid, Dr. med., University of Ulm
Other Study IDs: ULMNEONIRS04
Record Dates: First submitted 2011-09-06; First posted 2011-09-08 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Infant, Very Low Birth Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Very low birthweight infants

SUMMARY:
The purpose of this study is to examine the range of cerebral tissue oxygen saturation in healthy and sick very low birthweight infants during the first 72 hours of life.

DETAILED DESCRIPTION:
In this observational trial we want to examine cerebral tissue oxygen saturation, total hemoglobin, fractional tissue oxygen extraction and HbD as measured by near infrared spectroscopy during the first 72h of life in very low birthweight infants.

Differences between relatively healthy and sick preterm infants will be explored. A focus is to find differences between those infants who develop germinal matrix hemorrhage and those who are at risk only but do not develop hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Very low birthweight infants

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Very low birthweight infants treated in our hospital
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-04; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Cerebral tissue oxygen saturation during first 72 hours of life | during first 72 hours of life

CONTACTS AND LOCATIONS:
Overall Officials: Manuel B Schmid, Dr. med., Principal Investigator — University of Ulm
Locations (1):
- University Medical Center, Ulm, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Schwab AL, Mayer B, Bassler D, Hummler HD, Fuchs HW, Bryant MB. Cerebral Oxygenation in Preterm Infants Developing Cerebral Lesions. Front Pediatr. 2022 Apr 12;10:809248. doi: 10.3389/fped.2022.809248. eCollection 2022. PMID 35498781